CLINICAL TRIAL: NCT03727672
Title: Salivary Inflammatory Markers (Interleukin -1β, Interleukin -6, C- Reactive Protein) in Tension Type Headache and Migraine
Brief Title: Salivary Inflammatory Markers in Tension Type Headache and Migraine
Acronym: SalHead
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Anastasia Bougea, Clinical Researcher, National and Kapodistrian University of Athens
Other Study IDs: 638/5.11.2015
Record Dates: First submitted 2018-10-23; First posted 2018-11-01 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Migraine; Tension-Type Headache
Keywords: Primary headaches; CRP; Interleukin1β; Interleukin6; markers
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva transferrin levels were measured by competitive immunoassay kits and Interleukin-6, Interleukin-1β and CRP levels were measured by sandwich ELISA kits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tension type headache patients: 30 subjects of both genders, aged from 18 to 60 years old, with primary headaches (TTH) , according to the International Classification of Headache Disorders, 3rd edition (beta version) , were enrolled from the outpatient headache clinic of the first Neurological Hospital of University of Athens between January to March 2016.
- Migraine patients: 30 subjects of both genders, aged from 18 to 60 years old, with migraine, according to the International Classification of Headache Disorders, 3rd edition (beta version) , were enrolled from the outpatient headache clinic of the first Neurological Hospital of University of Athens between January to March 2016.
- age matched controls: 30 healthy control subjects aged matched were recruited mainly from hospital staff and patients' relatives

SUMMARY:
Data role of salivary inflammatory markers in migraine and Tension Type headache (TTH) are lacking. Τhe investigators studied whether headache attacks are associated with changes in C reactive protein (CRP), Interleukin -1β and Interleukin -6 in saliva in patients with Tension Type Headache and Migraine and age matched healthy controls . Τhe investigators, also investigated whether these markers could be influenced by comorbidities such as depression and anxiety.

DETAILED DESCRIPTION:
Sixty subjects of both genders, aged from 18 to 60 years old, with primary headaches TTH and migraine, according to the International Classification of Headache Disorders, 3rd edition (beta version), were enrolled from the outpatient headache clinic of University Hospital of Athens between January to March 2016. 30 healthy control subjects aged matched were recruited mainly from hospital staff and patients' relatives.

Initially, the participants completed the Hamilton Anxiety (HAM-A), Scale Beck Depression Inventory (BDI). All patients had to keep a headache diary during the four-week run-in period. All headache suffers were instructed to collected salivary headache-free baseline samples at the time of study screening when they had been free of headache for at least 48 hours (time point A). All headache suffers collected additional samples during moderate/severe headache (time point B), and at self-defined resolution phase 24 hours of their headache attack (time point C). Healthy control subjects were instructed to collected samples at the time of study screening (time point D). Every week, until four weeks and one month after the end of the study, participants were contacted, in order to ensure the compliance and the appropriate use of the technique. One year later longitudinal data would also be obtain.

Saliva Sample Collection Detailed instructions for the correct collection of saliva samples were given to all participants. Such instructions include avoiding eating a major meal and teeth brushing 60 minutes prior to sample collection. Also consumption of high sugar and caffeine content foods as well as high acidity foods have to be excluded before saliva sample collection. Mouth rinse with water in order to remove any food residue and saliva sample collection at least 10 minutes after mouth rinse was recommended. Unstimulated whole saliva that pooled on the mouth floor were collected from patients and healthy volunteers in high quality polypropylene vials by the passive drool technique. Finally, all samples were stored in a plastic container at 2-4 ° C until analysis. Saliva was collected from the participants, at 8.00 a.m. in the morning in order to rule out any confounding factor caused by circadian rhythm.

Sample Analysis Morning samples were kept in the refrigerator at 4°C and at the end of the day were brought to the laboratory where they were centrifuged 3000 rpm at 4°C and the supernatant was aliquoted in to polypropylene Cryogenic vials. Vials were frozen in -80°C until analyzed. Saliva transferrin levels were measured by competitive immunoassay kits and Interleukin-6, Interleukin-1β and CRP levels were measured by sandwich ELISA kits. Transferrin levels were used as a screening tool for the presence of blood in saliva samples and samples with transferrin values greater than 1 mg/dl were considered as candidates for exclusion in other salivary assays. Cortisol assay has a sensitivity of < 0.007 μg/ml and an inter-assay coefficient of variation of < 11% while these characteristics are 0.07 pg/ml and 8 for Interleukin-6, 0.37 pg/ml and 7 for Interleukin-1β, 10 pg/ml and 11.2 for CRP as well as 0.08 mg/dl and 7.2 for transferrin respectively.

ELIGIBILITY:
Inclusion Criteria:

* aged from 18 to 60 years old
* Tension type Headache (TTH) and migraine, fulfilling the criteria International Classification of Headache Disorders, 3rd edition (beta version)

Exclusion Criteria:

* abnormal plasma CRP, Interleukin-1β and Interleukin-6 levels (>10 mg/L)
* smoking cigarettes > 1 pack/day;
* current pregnancy, lactation, or hormonal contraceptive use
* alcohol or substance abuse
* drug use such as anticoagulants, statins, or hormonal drugs
* anti-inflammatory therapy
* other primary or secondary headaches
* major psychiatric disease
* oral health problems.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects of both genders, aged from 18 to 60 years old, with primary headaches TTH and migraine, according to the International Classification of Headache Disorders, 3rd edition (beta version), were enrolled from the outpatient headache clinic of the first Neurological Hospital of University of Athens between January to March 2016. Fifteen healthy control subjects aged matched were recruited mainly from hospital staff and patients' relatives
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
migraine/Tension type Headache and C reactive protein | 2 years
  establish whether attacks of migraine and Tension type Headache are associated with changes in the concentration of C reactive protein
migraine/Tension type Headache and Interleukin -1β | 2 years
  establish whether attacks of migraine and Tension type Headache are associated with changes in the concentration of Interleukin-1β
migraine/Tension type Headache and Interleukin-6 levels | 2 years
  establish whether attacks of migraine and Tension type Headache are associated with changes in the concentration of Interleukin-6 levels

SECONDARY OUTCOMES:
C reactive protein concentrations | 2 years
  C reactive protein concentrations as assessed using sandwich ELISA kits
Interleukin-1β concentrations | 2 years
  Interleukin-1β concentrations as assessed using sandwich ELISA kits
Interleukin-6 levels concentrations | 2,5 years
  Interleukin-6 levels concentrations as assessed using sandwich ELISA kits
Anxiety | 2,5 years
  Anxiety as assessed using the Hamilton Anxiety (HAM-A)
Depression | 2,5 years
  Depression as assessed using the Beck Depression Inventory (BDI)

CONTACTS AND LOCATIONS:
Overall Officials: ANASTASIA BOUGEA, PHD, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Eginition Hospital, National and Kapodistrian University of Athens, School of Medicine, Athens, Greece, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided
database

REFERENCES:
- [Result] Sjogren E, Leanderson P, Kristenson M, Ernerudh J. Interleukin-6 levels in relation to psychosocial factors: studies on serum, saliva, and in vitro production by blood mononuclear cells. Brain Behav Immun. 2006 May;20(3):270-8. doi: 10.1016/j.bbi.2005.08.001. Epub 2005 Sep 23. PMID 16183246